CLINICAL TRIAL: NCT01223027
Title: An Open-label, Randomized, Multi-center, Phase III Study to Compare the Safety and Efficacy of Dovitinib Versus Sorafenib in Patients With Metastatic Renal Cell Carcinoma After Failure of Anti-angiogenic (VEGF-targeted and mTOR Inhibitor) Therapies
Brief Title: Study of Dovitinib Versus Sorafenib in Patients With Metastatic Renal Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2302; 2009-015459-25 (EudraCT Number)
Record Dates: First submitted 2010-09-30; First posted 2010-10-18 (Estimated); Results first posted 2015-11-06 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-11

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Dovitinib; TKI; Renal cell cancer; RCC; mRCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dovitinib + best supportive care (BSC) (Experimental): Patients randomized to the dovitinib treatment arm received 500 mg of dovitinib orally on 5 days on/2 days off dosing schedule.
  Interventions: Drug: Dovitinib
- Sorafenib + BSC (Active Comparator): Patients in the sorafenib control arm received400 mg of sorafenib (2 x 200 mg tablets) orally taken twice daily.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Dovitinib — Dovitinib is formulated as an oral gelatin capsule of 100 mg strength and was dosed on a flat scale of 500 mg on a 5 days on/2 days off dosing schedule. Medication labels complied withthe legal requirements of each country and were printed in the local language.
  Other Names: TKI258
  Arms: Dovitinib + best supportive care (BSC)
Drug: Sorafenib — Sorafenib is formulated as a round, oral, biconvex, red film-coated tablet that contains 200 mg of sorafenib (tosylate). Sorafenib was administered twice daily without food at least 1 hour before or 2 hours after a meal. Sorafenib was supplied according to local practice.
  Arms: Sorafenib + BSC

SUMMARY:
This study will evaluate the safety and efficacy of Dovitinib versus sorafenib in patients with metastatic renal cell cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic renal cell carcinoma (mRCC) with histological or cytological confirmation of clear cell carcinoma or a component of clear cell
* Patients must have received one and only one prior VEGF-targeted therapy and one and only one prior mTOR inhibitor therapy in the metastatic setting. One VEGF targeted therapy (e.g. sunitinib, or pazopanib, or axitinib, or tivozanib or bevacizumab) and one prior mTOR inhibitor therapy (everolimus, or temsirolimus or ridaforolimus)
* Prior cytokines therapy and prior vaccines in the adjuvant setting is permitted.
* Patients must have had disease progression on or within 6 months of stopping the last therapy.
* Patients must have at least one measurable lesion at baseline (by RECIST Criteria Guidelines v1.1) assessed by Computer Tomography (CT) Scan or Magnetic Resonance Imaging (MRI).
* Karnofsky performance status ≥ 70%
* Patients must have the following laboratory values:

  * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hemoglobin (Hgb) > 9 g/dL
  * Serum total bilirubin: ≤ 1.5 x ULN
  * ALT and AST ≤ 3.0 x ULN (Patients with known liver metastases: AST and ALT ≤ 5.0 x ULN)
  * Serum creatinine ≤ 1.5 x ULN

Exclusion Criteria:

* Patients who have previously received sorafenib therapy in the neoadjuvant, adjuvant or metastatic setting.
* Patients who have previously received Dovitinib or brivanib in the neoadjuvant, adjuvant or metastatic setting.
* Patients with brain metastases. Radiological imaging (e.g. CT or MRI scan) of the brain is required at screening/baseline
* Patients with another primary malignancy within 3 years prior to starting study treatment, with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma or non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix
* Patients who have received the last administration of an anticancer targeted small molecule therapy ≤ 2 weeks prior to starting study treatment (e.g. sunitinib, pazopanib, axitinib, everolimus, temsirolimus), or who have not recovered from the side effects of such therapy
* Patients who have received the last administration of nitrosurea or mitomycin-C ≤ 6 weeks prior to starting study treatment, or who have not recovered from the side effects of such therapy
* Patients who have undergone major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) ≤ 4 weeks prior to starting study treatment or who have not recovered from side effects of such therapy
* Patients with a history of pulmonary embolism (PE), or untreated deep venous thrombosis (DVT) within the past 6 months
* Patients with concurrent severe and/or uncontrolled medical conditions which could compromise participation in the study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Actual)
Dates: Start 2011-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (179):
- United States (34):
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - University of California San Diego - Moores Cancer Center Dept of Moores Cancer Ctr (5), La Jolla, California
  - Cedars Sinai Medical Center Cedars Sinai Medical Ctr. (SC), Los Angeles, California
  - University of California at Los Angeles UCLA (4), Los Angeles, California
  - Stanford University Medical Center Cancer Clinical Trials Office, Stanford, California
  - Rocky Mountain Cancer Centers RMCC, Greenwood Village, Colorado
  - Florida Cancer Specialists DeptofFloridaCancerSpecialists, Fort Myers, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Straub Clinic & Hospital Straub, Honolulu, Hawaii
  - Moanalua Medical Center. Attn: Oncology Dept, Honolulu, Hawaii
  - University of Kansas Cancer Center Univ of KS, Kansas City, Kansas
  - University of Maryland Medical Center UMMC, Baltimore, Maryland
  - Karmanos Cancer Institute Dept.of KarmanosCancerInst (5), Detroit, Michigan
  - University of Minnesota Medical Center - Fairview Univ of MN, Minneapolis, Minnesota
  - Comprehensive Cancer Centers of Nevada CCC of Nevada (1), Las Vegas, Nevada
  - CINJ at Cooper University Hospital Cooper, Voorhees Township, New Jersey
  - Memorial Sloan Kettering Cancer Center Dept. of MSKCC, New York, New York
  - SUNY - Upstate Medical University Div. of Hematology-Oncology, Syracuse, New York
  - New York Oncology Hematology, P.C. Dept. of New York Oncology. PC, Troy, New York
  - Willamette Valley Clinical Studies Williamette Valley Cancer, Eugene, Oregon
  - St. Luke's Hospital and Health Network St Luke's, Bethlehem, Pennsylvania
  - Medical University of South Carolina -Hollings Cancer Center Med Univ SC, Charleston, South Carolina
  - Cancer Centers of the Carolinas CC of C -Eastside, Greenville, South Carolina
  - Sarah Cannon Research Institute SC - 3, Chattanooga, Tennessee
  - The West Clinic, Memphis, Tennessee
  - Vanderbilt University Medical Center SC, Nashville, Tennessee
  - Baylor Health Care System/Sammons Cancer Center Dept. of Sammons Cancer (4), Dallas, Texas
  - Texas Oncology Texas Onc - Austin, Dallas, Texas
  - Texas Oncology Texas Oncology - Houston, Dallas, Texas
  - University of Texas Southwestern Medical Center UTSW, Dallas, Texas
  - Deke Slayton Cancer Center Deke Slayton Cancer Center (2), Webster, Texas
  - Utah Cancer Specialists Dept.of Utah Cancer Spec. (3), Salt Lake City, Utah
  - University of Virginia Health Systems Univ Virginia, Charlottesville, Virginia
  - Rockwood Clinic Spokane Location, Spokane, Washington
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Rosario, Sante Fe
- Australia (6):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Woodville, South Australia
  - Novartis Investigative Site, Footscray, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
- Novartis Investigative Site, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (10):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Novartis Investigative Site, Bogotá, Colombia
- Czechia (3):
  - Novartis Investigative Site, Brno, Czech Republic
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- France (17):
  - Novartis Investigative Site, Suresnes, France
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Saint-Priest-en-Jarez
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandoeuvre-Les-Nancy Cede
  - Novartis Investigative Site, Villejuif
- Germany (16):
  - Novartis Investigative Site, Aschaffenburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Weiden
- Greece (3):
  - Novartis Investigative Site, Athens, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Szolnok
- Israel (3):
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Zrifin
- Italy (9):
  - Novartis Investigative Site, Arezzo, AR
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Napoli
- Japan (22):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Chiba, Chiba
  - Novartis Investigative Site, Tōon, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Hiroshima, Hiroshima
  - Novartis Investigative Site, Obihiro, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Sayama, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Hidaka, Saitama
  - Novartis Investigative Site, Kitaadachi-gun, Saitama
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Koto, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Yamagata, Yamagata
- Netherlands (6):
  - Novartis Investigative Site, Meerssen, KR
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Dordrecht
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Rotterdam
- Norway (2):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigative Site, Bergen
- Novartis Investigative Site, Warsaw, Poland
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Bratislava, Slovak Republic, Slovakia
- Novartis Investigative Site, Seoul, Korea, South Korea
- Spain (17):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Palma de Mallorca, Balearic Islands
  - Novartis Investigative Site, Barcelona, Barcelona
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Las Palmas de Gran Canarias, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Benidorm, Valencia
  - Novartis Investigative Site, Valencia, Valencia
- Sweden (4):
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Sundsvall
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Novartis Investigative Site, Bangkok, Thailand
- United Kingdom (7):
  - Novartis Investigative Site, Bristol, Avon
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Colchester
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Motzer RJ, Porta C, Vogelzang NJ, Sternberg CN, Szczylik C, Zolnierek J, Kollmannsberger C, Rha SY, Bjarnason GA, Melichar B, De Giorgi U, Grunwald V, Davis ID, Lee JL, Esteban E, Urbanowitz G, Cai C, Squires M, Marker M, Shi MM, Escudier B. Dovitinib versus sorafenib for third-line targeted treatment of patients with metastatic renal cell carcinoma: an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Mar;15(3):286-96. doi: 10.1016/S1470-2045(14)70030-0. Epub 2014 Feb 17. PMID 24556040

RESULTS

PARTICIPANT FLOW:
Groups:
- Dovitinib + Best Supportive Care (BSC): Patients randomized to the dovitinib treatment arm received 500 mg of dovitinib taken orally on 5 days on/2 days off dosing schedule.
- Sorafenib + BSC: Patients in the sorafenib control arm received 400 mg of sorafenib (2 x 200 mg tablets) taken orally twice daily.
Period: Overall Study
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Started | 284 | 286
Completed | 10 (Completed = Ongoing at data cut-off of 25-Jan-2013) | 9 (Completed = Ongoing at data cut-off of 25-Jan-2013)
Not Completed | 274 | 277
Not completed — Adverse Event | 20 | 10
Not completed — Death | 42 | 42
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 4 | 8
Not completed — Progressive Disease | 167 | 183
Not completed — Protocol Violation | 2 | 1
Not completed — Subject/guardian decicion | 18 | 16
Not completed — New therapy for study indication | 17 | 8
Not completed — Study terminated by sponsor | 2 | 8

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC | Total
Number analyzed (Participants) | 284 | 286 | 570
Age, Customized [Number; unit: Participants]
  < 65 years | 187 | 165 | 352
  >= 65 years | 97 | 121 | 218
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 67 | 138
  Male | 213 | 219 | 432
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 233 | 232 | 465
  Asian | 42 | 40 | 82
  Black | 3 | 5 | 8
  Unknown | 1 | 6 | 7
  Other | 5 | 3 | 8
Weight [Mean (Standard Deviation); unit: kg] | 74.9 (15.39) | 75.5 (15.96) | 75.2 (15.67)
Karnofsky performance score [Number; unit: Participants]
  100 -Normal no complaints; no evidence of disease | 83 | 73 | 156
  90 - Able to carry on normal activity | 93 | 101 | 194
  80 - Normal activity with efforts | 73 | 83 | 156
  70 - Cares for self | 35 | 29 | 64
Memorial Sloan Kettering Cancer Center Risk Criteria (MSKCC) risk group [Number; unit: Participants] — Pts were place into 3 distinct risk groups based on the number of risk factors that the patient had at baseline:
  Low Karnofsky Performance Status: <80%, Low serum hemoglobin: males (≤ 13 g/dL); females (≤ 11.5 g/dL), High corrected serum calcium: ≥ 10 mg/dL. Pts in the favorable group are expected to live longer while patients in the poor risk group are expected to die sooner than the patients in the other groups.
  Favorable = Pt. had none of the risks; Intermediate = Patient had 1 risk factor; Poor = Pt. had 2 or 3 risk factors Missing = not enough information at baseline to categorize
  Participants
    Favorable | 70 | 65 | 135
    Intermediate | 156 | 155 | 311
    Poor | 54 | 61 | 115
    Missing | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per Independent Central Radiology Review
Description: Assessed according to RECIST 1.1. PFS was defined as the time from the date of randomization to the date of the first documented disease progression or death due to any cause. If a patient had not progressed or died, on the date of the analysis cut-off or when he/she received any further anti-neoplastic therapy, PFS was censored on the date of last tumor assessment before the cutoff date or the anti-neoplastic therapy date. The distribution of PFS was estimated using the Kaplan-Meier method. The median PFS along with 95% confidence intervals was presented by treatment group.
Time Frame: Until disease progression or discontinuation of treatment due to unacceptable toxicity up to 30-Jun-2014 (discontinuation)
Population: Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Number analyzed (Participants) | 284 | 286
Months | 3.7 [3.5 to 3.9] | 3.6 [3.5 to 3.7]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was the key secondary endpoint and was defined as the time from date of randomization to the date of death due to any cause. If a patient was not known to have died, survival was censored on the date of last contact.
Time Frame: until at least 386 deaths are documented in the clinical database.
Population: Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Number analyzed (Participants) | 284 | 286
Months | 11.1 [9.5 to 13.4] | 11.0 [8.6 to 13.5]

3. Secondary Outcome: Progression Free Survival (PFS) Per Investigator's Radiology Review
Description: PFS was defined as the time from the date of randomization to the date of the first documented disease progression or death due to any cause. The primary analysis for PFS (based on central review) was also to be repeated on FAS considering the Investigator assessments and using the same analytical conventions as the primary analysis.
Time Frame: Until disease progression or discontinuation of treatment due to unacceptable toxicity
Population: Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Number analyzed (Participants) | 284 | 286
Months | 3.9 [3.7 to 5.1] | 3.9 [3.7 to 5.0]

4. Secondary Outcome: Percentage of Participants With Overall Response Rate (ORR) by Central Radiology Review
Description: Overall response rate (ORR) was defined as the proportion of patients with best overall response of complete response (CR) or partial response (PR). Best overall esponse (BOR) for each patient was determined from the sequence of overall (lesion) responses according to the following rules: CR = at least two determinations of CR at least 4 weeks apart before progression where confirmation required or one determination of CR prior to progression where confirmation not required. CR = at least two determinations of CR at least 4 weeks apart before progression where confirmation required or one determination of CR prior to progression where confirmation not required. SD = at least one SD assessment (or better) > 6 weeks after randomization (and not qualifying for CR or PR). PD = progression ≤ 17 weeks after randomization (and not qualifying for CR, PR or SD).
Time Frame: Until disease progression or discontinuation of treatment due to unacceptable toxicity
Population: Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Number; unit: Percentage of Participants
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Number analyzed (Participants) | 284 | 286
Percentage of Participants | 3.9 | 3.8

5. Secondary Outcome: Time to Definitive Worsening of Karnofsky Performance Status (KPS)
Description: Time to definitive worsening of Karnofsky performance status (KPS) was defined as the time from date of randomization to the date of definitive worsening of KPS or to the date of death whichever occurred earlier. Definitive worsening was defined as a definitive decrease in performance status by at least one Karnofsky category (i.e. at least 10 points less) compared to Baseline. Worsening was considered definitive if no later increase above the defined threshold was observed within the course of the study. A single measure reporting a decrease in Karnofsky performance status was sufficient to consider it as definitive only if it was the last one available for this patient. Time to definitive worsening of KPS was analyzed at the time of the final analysis for PFS.
Time Frame: from date of randomization to the date of definitive worsening of KPS or to the date of death whichever occurred earlier
Population: Full Analysis Set (FAS) consited of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Number analyzed (Participants) | 284 | 286
Months | 5.1 [3.8 to 6.5] | 5.7 [4.6 to 7.4]

6. Secondary Outcome: Patient-reported Outcomes (PROs): Time to Deterioration of Functional Assessment of Cancer Therapy-Kidney Symptom Index, Disease Related Symptoms (FKSI-DRS) by at Least 2 Scores
Description: The Kidney Cancer Symptom Index - Disease Related Symptoms (FKSI-DRS) is a validated symptom scale used in studies of patients with kidney cancer. It includes 9-items that assess pain, bone pain, fatigue, lack of energy, shortness of breath, fevers, weight loss, coughing, and blood in urine and responses to each question are answered on a 5-point Likert-type scale ranging from 0 to 4 (e.g., 0 = not at all; 1 = a little bit; 2 = somewhat; 3 = quite a bit; 4 = very much). FKSI-DRS scores range from 0 to 36, where higher scores correspond to better outcomes (eg, fewer symptoms).
Time Frame: from date of randomization, at least 2 score units
Population: Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Number analyzed (Participants) | 284 | 286
Months | 4.9 [4.5 to 6.6] | 6.4 [5.5 to 7.7]

7. Secondary Outcome: Patient-reported Outcomes (PROs): Time to Definitive Deterioration of the Physical Functioning (PF) Scale of EORTC QLQ-C30 by at Least 10%
Description: The EORTC QLQ-C30 contains 30 items and is composed of both multi-item scales and single-item measures. These include five functional scales (physical, role, emotional, social and cognitive functioning), three symptom scales (fatigue, pain, nausea, and vomiting), a global health status/QoL scale, and six single items (dyspnea, diarrhea, constipation, anorexia, insomnia and financial impact). Each of the multiitem scales includes a different set of items - no item occurs in more than one scale. Each item in the EORTC QLQ-C30 has 4 response categories (1=Not at all, 2= A little, 3= Quite a bit, 4= Very much) with the higher number representing a worse outcome.
Time Frame: from date of randomization
Population: Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Number analyzed (Participants) | 284 | 286
Months | 3.8 [3.2 to 4.6] | 5.6 [4.5 to 6.4]

8. Secondary Outcome: Patient-reported Outcomes (PROs): Time to Definitive Deterioration of the Quality of Life (QoL) Scale Scores of EORTC QLQ-C30 by at Least 10%
Description: as for outcome 7
Time Frame: from date of randomization
Population: Full Analysis Set (FAS) consisted of all randomized patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dovitinib + Best Supportive Care (BSC) | Sorafenib + BSC
Number analyzed (Participants) | 284 | 286
Months | 3.7 [2.8 to 4.6] | 4.5 [3.7 to 5.5]

9. Secondary Outcome: Pre-dose Concentration in Plasma in Dovitinib
Description: Predose concentrations of dovitinib were summarized by visit using PAS. All concentration data was listed by patient and time point using FAS. Mean pre-dose concentrations along with standard deviation (SD) was plotted over time if appropriate.
Time Frame: Week 2 Day 5, Week 4 Day 5, Week 6 Day 5
Population: Pharmacokinetic Analysis Set (PAS) consisted of all patients who received at least one dose of dovitinib and had at least one evaluable post-Baseline dovitinib concentration measurement.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dovitinib + Best Supportive Care (BSC)
Number analyzed (Participants) | 284
ng/ml
  Week 2 Day 5 (n: 205) | 128.06 (92.571)
  Week 4 Day 5 (n: 202) | 114.08 (77.884)
  Week 6 Day 5 (n: 170) | 118.27 (84.246)

ADVERSE EVENTS:
Description: 570 patients randomized, 564 patients included in the Safety Set. AEs were reported based on this set which consisted of all patients who received at least 1 dose of study treatment. Patients were analyzed according to treatment actually received which was defined as the treatment the patient received at the first day of study medication.
Groups:
- Dovitinib: Patients randomized to the dovitinib treatment arm received 500 mg of dovitinib taken orally on 5 days on/2 days off dosing schedule.
- Sorafenib: Patients in the sorafenib control arm received 400 mg of sorafenib (2 x 200 mg tablets) taken orally twice daily.
Arm/Group | Dovitinib | Sorafenib
Serious Adverse Events (participants affected / at risk) | 133/280 | 112/284
Other Adverse Events (participants affected / at risk) | 268/280 | 271/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dovitinib (N=280) | Sorafenib (N=284)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 | 0
CARDIAC TAMPONADE (Cardiac disorders) | 1 | 0
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 1
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 1 | 0
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 2
TACHYCARDIA (Cardiac disorders) | 1 | 0
HYPERCALCAEMIA OF MALIGNANCY (Endocrine disorders) | 0 | 1
DIPLOPIA (Eye disorders) | 1 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 7 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 | 2
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 | 1
ANAL FISSURE (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 2
COLONIC FISTULA (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 2
DIARRHOEA (Gastrointestinal disorders) | 10 | 4
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 3 | 0
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 | 0
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL MOTILITY DISORDER (Gastrointestinal disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 2 | 2
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 | 0
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 1 | 0
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 3
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 0 | 3
ODYNOPHAGIA (Gastrointestinal disorders) | 0 | 1
ORAL PAIN (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 2 | 0
PNEUMOPERITONEUM (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 | 1
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 3
VOMITING (Gastrointestinal disorders) | 8 | 3
ASTHENIA (General disorders) | 3 | 6
DEATH (General disorders) | 1 | 0
FATIGUE (General disorders) | 4 | 5
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 7 | 14
MALAISE (General disorders) | 2 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 1 | 0
PAIN (General disorders) | 3 | 3
PERFORMANCE STATUS DECREASED (General disorders) | 1 | 3
PYREXIA (General disorders) | 7 | 5
SUDDEN DEATH (General disorders) | 0 | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 1
JAUNDICE CHOLESTATIC (Hepatobiliary disorders) | 1 | 0
SERUM SICKNESS (Immune system disorders) | 1 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 1
CYSTITIS (Infections and infestations) | 1 | 0
EMPHYSEMATOUS CYSTITIS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 1
INFECTIVE GLOSSITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 7 | 8
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 4
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 1 | 0
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 | 1
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 | 1
AMYOTROPHY (Musculoskeletal and connective tissue disorders) | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 7
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEONECROSIS OF JAW (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 2
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
METASTATIC PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
APHASIA (Nervous system disorders) | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 2 | 0
DEPRESSED LEVEL OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 0
EPILEPSY (Nervous system disorders) | 1 | 0
HEMIPARESIS (Nervous system disorders) | 1 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0
NEURALGIA (Nervous system disorders) | 1 | 0
NEUROLOGICAL DECOMPENSATION (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 1
PRESYNCOPE (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
SPINAL CORD COMPRESSION (Nervous system disorders) | 2 | 2
SYNCOPE (Nervous system disorders) | 2 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
APATHY (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 3 | 2
DELIRIUM (Psychiatric disorders) | 1 | 0
AZOTAEMIA (Renal and urinary disorders) | 2 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 3
POLLAKIURIA (Renal and urinary disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
URINARY BLADDER HAEMORRHAGE (Renal and urinary disorders) | 0 | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0
URINARY RETENTION (Renal and urinary disorders) | 1 | 1
GENITAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 | 1
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
BRONCHIAL OBSTRUCTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 16 | 15
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 10 | 10
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 | 3
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 1
DIABETIC FOOT (Skin and subcutaneous tissue disorders) | 0 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 | 1
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 0
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0
SKIN LESION (Skin and subcutaneous tissue disorders) | 0 | 1
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 0 | 1
TOXIC SKIN ERUPTION (Skin and subcutaneous tissue disorders) | 0 | 1
EMBOLISM (Vascular disorders) | 2 | 0
HYPERTENSION (Vascular disorders) | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 2
PHLEBITIS (Vascular disorders) | 1 | 0
SHOCK (Vascular disorders) | 1 | 0
THROMBOSIS (Vascular disorders) | 1 | 0
VASCULAR FRAGILITY (Vascular disorders) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 7 | 7
LEUKOPENIA (Blood and lymphatic system disorders) | 2 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 1 | 0
GENERALISED OEDEMA (General disorders) | 2 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 1 | 1
MENINGITIS CRYPTOCOCCAL (Infections and infestations) | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 7 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 2
CONTRAST MEDIA REACTION (Injury, poisoning and procedural complications) | 1 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
AMYLASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 0 | 1
HAEMATOCRIT DECREASED (Investigations) | 0 | 1
LIPASE INCREASED (Investigations) | 1 | 0
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1
PLATELET COUNT DECREASED (Investigations) | 2 | 0
TROPONIN INCREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 2 | 0
CACHEXIA (Metabolism and nutrition disorders) | 2 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 4
DEHYDRATION (Metabolism and nutrition disorders) | 6 | 5
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 3 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 2
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOPHAGIA (Metabolism and nutrition disorders) | 2 | 0
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 1 | 0
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
EPIDURITIS (Nervous system disorders) | 1 | 0
HYDROPNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dovitinib (N=280) | Sorafenib (N=284)
ANAEMIA (Blood and lymphatic system disorders) | 27 | 28
HYPOTHYROIDISM (Endocrine disorders) | 14 | 8
LACRIMATION INCREASED (Eye disorders) | 19 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 34 | 37
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 28 | 23
CONSTIPATION (Gastrointestinal disorders) | 49 | 67
DIARRHOEA (Gastrointestinal disorders) | 184 | 126
DRY MOUTH (Gastrointestinal disorders) | 23 | 12
DYSPEPSIA (Gastrointestinal disorders) | 30 | 14
NAUSEA (Gastrointestinal disorders) | 146 | 81
STOMATITIS (Gastrointestinal disorders) | 31 | 53
VOMITING (Gastrointestinal disorders) | 120 | 44
ASTHENIA (General disorders) | 63 | 44
FATIGUE (General disorders) | 113 | 94
NON-CARDIAC CHEST PAIN (General disorders) | 22 | 18
OEDEMA PERIPHERAL (General disorders) | 26 | 17
PYREXIA (General disorders) | 40 | 37
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 25 | 5
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 25 | 8
LIPASE INCREASED (Investigations) | 16 | 11
WEIGHT DECREASED (Investigations) | 61 | 87
DECREASED APPETITE (Metabolism and nutrition disorders) | 90 | 96
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 55 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 26 | 26
BACK PAIN (Musculoskeletal and connective tissue disorders) | 37 | 32
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 18 | 24
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 15 | 6
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 15 | 13
MYALGIA (Musculoskeletal and connective tissue disorders) | 27 | 17
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 35 | 29
DIZZINESS (Nervous system disorders) | 27 | 7
DYSGEUSIA (Nervous system disorders) | 31 | 8
HEADACHE (Nervous system disorders) | 26 | 24
INSOMNIA (Psychiatric disorders) | 15 | 19
COUGH (Respiratory, thoracic and mediastinal disorders) | 50 | 48
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 22 | 25
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 51 | 48
ALOPECIA (Skin and subcutaneous tissue disorders) | 2 | 61
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 23 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 22 | 26
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 15
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 32 | 114
PRURITUS (Skin and subcutaneous tissue disorders) | 15 | 30
RASH (Skin and subcutaneous tissue disorders) | 54 | 47
HYPERTENSION (Vascular disorders) | 54 | 78

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.